CLINICAL TRIAL: NCT02907957
Title: A Clinical Evaluation Of Infrared Thermography To Assess Successful Caudal Block In Children
Brief Title: Infrared Thermography for Assessment of Caudal Block in Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ann & Robert H Lurie Children's Hospital of Chicago (Other)
Responsible Party: Principal Investigator, Luis Sequera-Ramos, Resident Physician, Anesthesiology, Ann & Robert H Lurie Children's Hospital of Chicago
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: IRB 2016-590
Record Dates: First submitted 2016-09-09; First posted 2016-09-20 (Estimated); Last update posted 2019-08-20 (Actual); Status verified 2018-07

CONDITIONS: Anesthesia, Conduction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Caudal (Active Comparator): Participants receiving a caudal neuraxial blockade, as clinically indicated.
  Interventions: Device: FLIR ONE; Procedure: Regional Anesthesia - Caudal Nerve Block
- No Caudal (Sham Comparator): Participants not receiving a caudal neuraxial blockade, as clinically indicated.
  Interventions: Device: FLIR ONE

INTERVENTIONS:
Device: FLIR ONE — Thermographic assessment of the lower extremities is obtained using the FLIR ONE smartphone camera and software.
Procedure: Regional Anesthesia - Caudal Nerve Block — Nerve block placement as a pain management strategy indicated for certain urological and lower extremity surgeries.
  Arms: Caudal

SUMMARY:
Regional analgesia via caudal neuraxial blockade provides pain relief for pediatric patients following urological and lower extremity procedures. The injection of local anesthetic into the caudal epidural space causes a sensory loss. This sympathetic blockade in turn causes a vasodilation, or increased blood flow, to the lower extremities.

The purpose of this study is to determine whether the FLIR ONE thermographic camera, a smartphone attachment which utilizes an application ("app") to measure the temperature at a site on an image of the lower extremity, will be able to differentiate between caudal, non-caudal, and failed caudal images.

ELIGIBILITY:
Inclusion Criteria:

* Children from 6mos to 5 years of age requiring general anesthesia and a caudal block for a surgical procedure

Exclusion Criteria:

* Patients with preexisting conditions that could affect the skin temperature on the lower extremities such as infection, edema, vascular disorder, etc.
* American Society of Anesthesiologists comorbidity ranking of 4 or greater
* Patient with contraindications for a caudal block such as: history of allergic, reactions to local anesthetics, coagulopathy, infection at the injection site, spinal abnormality, peripheral neurological disease, Raynaud's disease

Ages: 6 Months to 5 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 14 (Actual)
Dates: Start 2016-09 (Actual); Primary Completion 2018-06 (Actual); Study Completion 2018-06-28 (Actual)

PRIMARY OUTCOMES:
Predictive value of FLIR ONE | Assessments will be done through study completion, an average of 1 week following procedure.
  Reviewers blinded to intervention groups will asses patient pre-caudal, 1, 2, 3, 4, and 5 minute post-caudal images and rate whether, based on the image, they believe the patient received a caudal or not. The sensitivity and specificity of the FLIR ONE as a diagnositic tol will then be determined.

SECONDARY OUTCOMES:
Inter- and Intra- rater reliability | Assessments will be done through study completion, an average of 1 week following procedure.
  Reviewers will evaluate patient image at two separate ties at least a week apart. Recorded images will be compared within and between reviewers.
Temperature differences between pre-caudal and 5 minute post-caudal images | Images will be captured prior to caudal and 5 minutes immediately afterwards. Assessments will be done through study completion, an average of 1 week following procedure.
  Temperature differences between pre-caudal and 5 minute images will be summarized in both groups. Images in the non-caudal group will be taken at similar time points following anesthesia induction relative to caudal group patients.

CONTACTS AND LOCATIONS:
Overall Officials: Luis Sequera-Ramos, MD, Principal Investigator — Ann & Robert H Lurie Children's Hospital of Chicago
Locations (1):
- Ann & Robert H. Lurie Children's Hospital, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Suresh S, Long J, Birmingham PK, De Oliveira GS Jr. Are caudal blocks for pain control safe in children? an analysis of 18,650 caudal blocks from the Pediatric Regional Anesthesia Network (PRAN) database. Anesth Analg. 2015 Jan;120(1):151-156. doi: 10.1213/ANE.0000000000000446. PMID 25393589